CLINICAL TRIAL: NCT02470455
Title: Effect of Atorvastatin on Glycemic Control in Prediabetic Patients
Status: Completed | Type: Observational
Sponsor: Shri Ramachandra Bhanj Medical College (Other)
Responsible Party: Principal Investigator, Dr. Sansita Parida, Resident, Shri Ramachandra Bhanj Medical College
Other Study IDs: IEC/SCB/Pharma/2011/05
Record Dates: First submitted 2015-06-04; First posted 2015-06-12 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Prediabetic State
Keywords: Atorvastatin; Prediabetics; HbA1c
MeSH Terms: conditions — Prediabetic State | interventions — Atorvastatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Normoglycemic group: 25 patients were recruited who were on Atorvastatin and with normal blood glucose and Hb1Ac level.
  Interventions: Drug: Atorvastatin
- Prediabetic with normal GTT: 25 patients were recruited who were on Atorvastatin and with fasting blood sugar level 100-125 mg/dl with normal GTT.
  Interventions: Drug: Atorvastatin
- Prediabetic with impaired GTT: 25 patients were recruited who were on Atorvastatin and with fasting blood sugar level 100-125 mg/dl with impaired GTT.
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Some patients were receiving 20 mg of Atorvastatin wheras others were on a higher dose of 40-80mg daily. Patients were taking statins for either dyslipidemia, or primary or secondary prevention of cardiovascular disease.

SUMMARY:
The study was conducted to find out any possible effect of Atorvastatin on glycemic parameters in prediabetic patients.

DETAILED DESCRIPTION:
Diabetes is a growing public health problem throughout the world, threatening global health and economic prosperity. Currently, approximately 171 to 194 million people in the world have diabetes, the majority of the cases being Type II. This number is expected to increase to more than 330 million by the year 2025-a record doubling within a single generation. India with 62.2 million diabetic patients is fast becoming the diabetes capital of the world with possibility of the number of diabetic patients reaching the 80 million mark by 2030. Every sixth diabetic in the world is an Indian. China with 43.2 million patients comes second, followed by the US where 26.8 million people suffer from the disease.

This spectacular increase in the frequency of Type II diabetes is being paralleled by a similarly alarming increase in obesity, which is one of the major risk factors for Type II diabetes. Because of the close linkage of these two conditions, Ziv and Shafrir have suggested the term "diabesity" to describe this association. This dual epidemic which was largely ignored by the public health community until recently has come as a great surprise involving enormous economic burden as well as in terms of health. Disorders of glucose metabolism are associated with increased risk for cardiovascular disease (CVD) complications, including coronary, peripheral and cerebral arterial disease, that account for the majority of morbidity and mortality among patients with diabetes mellitus (DM).

Type II diabetes is commonly associated with dyslipidaemia, which represents a synergistic risk factor for cardiovascular disease. The National Cholesterol Education Program Adult Treatment Panel III (ATP III) listed diabetes as a coronary heart disease (CHD) risk equivalent for setting therapeutic goals for LDL cholesterol. A goal for LDL cholesterol of <100 mg/dl was recommended for patients with CHD and CHD risk equivalents. For the majority of patients with diabetes, this LDL cholesterol goal would evoke the use of cholesterol-lowering drugs, particularly statins. Some Interventional studies emphasized that statin treatment leads to a reduction in cardiovascular events independent of lipid reduction with possible benefits for patients with Type II diabetes. Statins could also contribute to diabetes prevention owing to lipid-lowering and so-called pleiotropic action. Statins improve endothelial function, inhibit smooth muscle cell proliferation, and reduce oxidative stress and inflammation. Thus, with recent FDA approved indications for statins being widened, statins are currently amongst the most widely used drugs in patients with or without diabetes.

Although statin therapy reduces cardiovascular risk, its relationship with the development of diabetes is controversial. Retrospective analysis of the West of Scotland Coronary Prevention Study (WOSCOPS) revealed that 5 years of treatment with pravastatin reduced diabetes incidence by 30%. The authors suggested that although lowering of triglyceride levels could influence diabetes incidence, other mechanisms such as anti-inflammatory action may be involved. On the contrary, pravastatin did not decrease diabetes incidence in another trial including glucose-intolerant humans, suggesting that early inception of statin therapy may be required for effective diabetes prevention. Likewise, simvastatin did not affect diabetes incidence in patients with atherosclerosis in the Heart Protection Study. In contrast, atorvastatin marginally increased diabetes incidence in the Anglo-Scandinavian Cardiac Outcomes Trial (ASCOT-LLA), which could be explained by statistical variation.

A recent review of 13 studies by Naveed Sattar, et al. published in The Lancet in 2010, on statins and their side-effects including a total of more than 91,140 participants suggested that use of statins is associated with increased risk of Type II diabetes by 9%.

However researchers of this meta-analysis have stressed that this study does not prove that statins directly raise the risk of Type II diabetes, but it raises the possibility of either a direct or indirect link between statins and diabetes that merits further investigation. Thus, exploring the role of statins in the initiation or progression of diabetes mellitus is an exciting area for investigation.

ELIGIBILITY:
Inclusion Criteria:

* Any patient on statins therapy whose blood sugar level is within normal limit.
* Pre-diabetic patients (IFG and/or IGT) on statins
* Patients who agreed to participate in the study and signed the informed consent form without any external motivation

Exclusion Criteria:

* Diagnosed cases of DM, both type I and II, on different anti-diabetic regimen
* Patients on β-blockers, thiazide diuretics, corticosteroids, which can affect blood sugar level
* Pregnancy and lactation
* Co-existing or other organ involvement like kidney, liver which can affect blood sugar level

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population was selected from patients attending Cardiology and Medicine Outpatient Department of S.C.B. Medical College, Cuttack, following inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2011-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in Glycosylated Hemoglobin (HbA1c) from baseline | At baseline and at 6 monhts, 12 months and 18 months follow up

SECONDARY OUTCOMES:
Change in Fasting blood sugar from baseline | At baseline and at 6 monhts, 12 months and 18 months follow up
Change in Post prandial blood sugar from baseline | At baseline and at 6 monhts, 12 months and 18 months follow up
Lipid profile | At baseline

CONTACTS AND LOCATIONS:
Overall Officials: TRUPTI R SWAIN, MD, Study Director — SCB Medical College, Cuttack, Odisha
Locations (1):
- SCB Medical College, Cuttack, Odisha, India

REFERENCES:
- [Result] Cholesterol Treatment Trialists' (CTT) Collaborators; Kearney PM, Blackwell L, Collins R, Keech A, Simes J, Peto R, Armitage J, Baigent C. Efficacy of cholesterol-lowering therapy in 18,686 people with diabetes in 14 randomised trials of statins: a meta-analysis. Lancet. 2008 Jan 12;371(9607):117-25. doi: 10.1016/S0140-6736(08)60104-X. PMID 18191683
- [Result] Forrester JS, Libby P. The inflammation hypothesis and its potential relevance to statin therapy. Am J Cardiol. 2007 Mar 1;99(5):732-8. doi: 10.1016/j.amjcard.2006.09.125. Epub 2007 Jan 10. PMID 17317382
- [Result] Freeman DJ, Norrie J, Sattar N, Neely RD, Cobbe SM, Ford I, Isles C, Lorimer AR, Macfarlane PW, McKillop JH, Packard CJ, Shepherd J, Gaw A. Pravastatin and the development of diabetes mellitus: evidence for a protective treatment effect in the West of Scotland Coronary Prevention Study. Circulation. 2001 Jan 23;103(3):357-62. doi: 10.1161/01.cir.103.3.357. PMID 11157685
- [Result] Keech A, Colquhoun D, Best J, Kirby A, Simes RJ, Hunt D, Hague W, Beller E, Arulchelvam M, Baker J, Tonkin A; LIPID Study Group. Secondary prevention of cardiovascular events with long-term pravastatin in patients with diabetes or impaired fasting glucose: results from the LIPID trial. Diabetes Care. 2003 Oct;26(10):2713-21. doi: 10.2337/diacare.26.10.2713. PMID 14514569
- [Result] Sattar N, Preiss D, Murray HM, Welsh P, Buckley BM, de Craen AJ, Seshasai SR, McMurray JJ, Freeman DJ, Jukema JW, Macfarlane PW, Packard CJ, Stott DJ, Westendorp RG, Shepherd J, Davis BR, Pressel SL, Marchioli R, Marfisi RM, Maggioni AP, Tavazzi L, Tognoni G, Kjekshus J, Pedersen TR, Cook TJ, Gotto AM, Clearfield MB, Downs JR, Nakamura H, Ohashi Y, Mizuno K, Ray KK, Ford I. Statins and risk of incident diabetes: a collaborative meta-analysis of randomised statin trials. Lancet. 2010 Feb 27;375(9716):735-42. doi: 10.1016/S0140-6736(09)61965-6. Epub 2010 Feb 16. PMID 20167359
- [Result] Fisslthaler B, Michaelis UR, Randriamboavonjy V, Busse R, Fleming I. Cytochrome P450 epoxygenases and vascular tone: novel role for HMG-CoA reductase inhibitors in the regulation of CYP 2C expression. Biochim Biophys Acta. 2003 Feb 17;1619(3):332-9. doi: 10.1016/s0304-4165(02)00492-0. PMID 12573493
- [Result] Moosmann B, Behl C. Selenoprotein synthesis and side-effects of statins. Lancet. 2004 Mar 13;363(9412):892-4. doi: 10.1016/S0140-6736(04)15739-5. PMID 15031036